CLINICAL TRIAL: NCT05421585
Title: Comparison of the Effectiveness of Ultrasound-Guided Quadratus Lumborum 2 Block and Classic Thoracolumbar Interfacial Plane Block in the Management of Postoperative Analgesia After Lumbar Spinal Surgery
Brief Title: Comparison of the Effectiveness of Two Different Block in the Management of Postoperative Analgesia After Lumbar Spinal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun University (Other)
Responsible Party: Principal Investigator, Senay Canikli, medical specialist (Anesthesiology and Reanimation), Samsun University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 22-AKD-26
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: The Effect of Two Different Block Methods on Postoperative Pain Management in Lumbar Spinal Surgery
Keywords: Lumbar spinal surgery; Postoperative pain; QL2 block; TLIP block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: prospective randomized trial
Who Masked: Participant
Masking Description: Before coming to the operating room, the patients will be randomly divided into 2 groups (Group Q= QL2 block group, Group T= Classic TLIP group) each containing 26 patients, using a closed envelope method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QL2 block (Active Comparator): Posterior QLB process After aseptic conditions are provided, the convex US probe will be covered with a sterile sheath, and an 80-100 mm block needle will be used. After imaging the abdominal muscles with the anterior approach, the needle will be advanced in the Petit triangle and 1-2 ml of saline will be injected into the posterior border of the quadratus lumborum muscle. After the block location is confirmed, 20 ml of local anesthetic infiltration at a concentration of 0.25% will be applied. The same procedure will be applied to the other side. A total of 30 ml of local anesthetic solution will be used.
  Interventions: Other: observational drug study
- TLIP block (Active Comparator): Classic TLIP block After providing aseptic conditions, the high frequency linear US probe will be covered with a sterile sheath, and a 50 mm block needle will be used. The ultrasound probe will be placed vertically at the level of the L3 vertebra. After visualizing the guiding point spinous process and interspinal muscles, the probe will be moved laterally to visualize the longissimus and multifidus muscles. By using the in-plane technique, the block needle will be directed from medial to lateral, and after reaching the interfacial area between the longissimus and multifidus muscles, the block area will be confirmed by administering 5 ml of serum physiologically. Then, 20 ml of 0.25% local anesthetic will be administered. The same procedure will be applied to the other side. A total of 40 ml of local anesthetic solution will be used.
  Interventions: Other: observational drug study

INTERVENTIONS:
Other: observational drug study — Postoperative opioid consumption will be evaluated by applying 2 different block methods to patients who have undergone lumbar disc surgery

SUMMARY:
Lumbar spinal surgery, one of the most common operations for the treatment of back and leg pain, is a painful postoperative procedure. Pain control is an important part of the treatment in these patients who may develop chronic pain. In patients undergoing surgery for lumbar disc herniation (LDH), severe pain may occur in the postoperative period, especially in the operation area, and this pain may become chronic. The subject of our study is to observe the effect on the use of analgesics by randomizing the patients that we routinely block in this painful procedure. We aimed to evaluate the analgesic efficacy of two different regional analgesia methods performed under ultrasound guidance in patients undergoing lumbar spinal surgery.Thoracolumbar interfacial plane (TLIP) block is a regional analgesia technique performed under US guidance, which was defined by Hand et al. in 2015 (10). Ueshima et al. retrospectively demonstrated that this technique produces effective analgesia after lumbar laminoplasty.

reported in their study (11). In the classical technique, local anesthetic infiltration is performed between the Multifidus and Longissimus muscles in the 4th Lumbar (L4) vertebral region (10). There is no study in the literature comparing classical TLIP block and QL2 block.

In this study, it was aimed to compare the effectiveness of US-guided Classic TLIP block and Posterior QLB (QL2) block for postoperative analgesia management after LDH surgery. Our primary aim is to determine the 24-hour opioid requirement, and our secondary aim is to; to compare postoperative pain scores (NRS), to evaluate side effects (allergic reaction, nausea, vomiting) associated with opioid use and complications that may occur due to block.

DETAILED DESCRIPTION:
Objective: The aim of this study was to compare the efficacy of US-guided Classic TLIP block and Posterior QLB (QL2) block for postoperative analgesia management after LDH surgery. Our primary aim is to determine the 24-hour opioid requirement, and our secondary aim is to; compare postoperative pain scores (NRS), to evaluate side effects (allergic reaction, nausea, vomiting) associated with opioid use and complications that may occur due to block.

Content: Lumbar spinal surgery is one of the most common operations performed for the treatment of back and leg pain (1). Pain control is an important part of the treatment in these patients who may develop chronic pain. In patients undergoing surgery for lumbar disc herniation (LDH), severe pain may occur in the postoperative period, especially in the operation area, and this pain may become chronic (2). Effective postoperative pain control reduces complications such as hospital-acquired opioids are widely used analgesic agents. Parenteral opioids are preferred for the treatment of acute postoperative pain in most patients who have surgery. Although opioids are widely used in the treatment of acute postoperative pain. They may cause opioid-related adverse events (ORAE) such as nausea, vomiting, allergic reactions, sedation, and respiratory depression (3). In order to reduce the use of systemic opioids, regional anesthesia techniques may be preferred with the increase in the use of ultrasound (US) in daily anesthesia practice (4).

Quadratus lumborum block (QLB) performed under US guidance is an interfacial plane block defined by Blanco (5). This block is used in the management of analgesia after abdominal and lumbar surgery (5-9). Local anesthetic solution is injected around the quadratus lumborum muscle to block the thoracolumbar nerves. In posterior OLB (QL2) block, local anesthetic solution is injected from the posterior part of the muscle and spreads between the Quadratus lumborum and Erector spina muscles (6). Since it is performed under US guidance, it is an easy and reliable method with a low complication rate. and thromboembolism, as it provides early mobilization and early discharge.Thoracolumbar interfacial plane (TLIP) block is a regional analgesia technique performed under US guidance, which was defined by Hand et al. in 2015 (10). Ueshima et al. retrospectively demonstrated that this technique produces effective analgesia after lumbar laminoplasty.

reported in their study (11). In the classical technique, local anesthetic infiltration is performed between the Multifidus and Longissimus muscles in the 4th Lumbar (L4) vertebral region (10). There is no study in the literature comparing classical TLIP block and QL2 block.

In this study, it was aimed to compare the effectiveness of US-guided Classic TLIP block and Posterior QLB (QL2) block for postoperative analgesia management after LDH surgery. Our primary aim is to determine the 24-hour opioid requirement, and our secondary aim is to; to compare postoperative pain scores (NRS), to evaluate side effects (allergic reaction, nausea, vomiting) associated with opioid use and complications that may occur due to block Material and Method Sixty patients with ASA classification I-II, aged 18-65 years, scheduled for lumbar discectomy + laminectomy under general anesthesia will be included in this prospective, randomized study. Patients with a history of bleeding diathesis, taking anticoagulant therapy, allergic or sensitive to local anesthetic and opioid drugs, patients with infection in the area to be blocked, patients who have had previous lumbar surgery, patients using gabapentinoids or corticosteroids, patients who cannot use a patient-controlled anesthesia device, patients with suspected pregnancy , pregnant or lactating mothers and patients who do not accept the procedure will be excluded from the study.

1. General anesthesia After the patients are taken to the operating room, all patients will be premedicated with 2 mg of intravenous midazolam. In anesthesia induction, 2-2.5 mg kg-1 iv propofol, 1-1.5 mcg kg-1 iv fentanyl, 0.6 mg kg-1 iv rocuronium will be intubated. The patient will then be placed in the prone position. Anesthesia will be maintained with 1-2% sevoflurane and 50 mcg/hour remifentanil in a 50% oxygen-air mixture. Mechanical ventilator settings will be adjusted so that tidal volume is 6-8 ml/kg, maximum airway pressure is 30 cmH2 O, end tidal CO2 is 30-35mmHg. If the pulse or mean blood pressure increases by 20% from the preoperative value, a bolus of 25 mcg fentanyl and 0.1 mg kg-1 rocuronium will be administered. Lumbar discectomy + laminectomy will be performed by the same surgical team with the same routine surgical procedure. Patients will receive an analgesic regimen as described post-induction and pre-extubation. To prevent nausea and vomiting, iv 4 mg of ondansetron will be given. Patients with adequate spontaneous breathing will be taken to the postoperative recovery unit after extubating. Patients who reach 12 points in Aldrete scoring will be sent to the service. Before coming to the operating room, the patients will be randomly divided into 2 groups (Group Q= QL2 block group, Group T= Classic TLIP group) each containing 26 patients, using a sealed envelope method.
2. Block technique The block that we use routinely, in accordance with the guidelines and valid, will be applied to the patient in the preoperative block room 30 minutes before the operation starts (5-9).

   1. Posterior QLB process; After aseptic conditions are provided, the convex US probe will be covered with a sterile sheath, and an 80-100 mm block needle will be used. After imaging the abdominal muscles with the anterior approach, the needle will be advanced in the Petit triangle and 1-2 ml of saline will be injected into the posterior border of the quadratus lumborum muscle. After the block location is confirmed, 20 ml of local anesthetic infiltration at a concentration of 0.25% will be applied. The same procedure will be applied to the other side. A total of 30 ml of local anesthetic solution will be used.
   2. Classic TLIP block: Operation after providing aseptic conditions, the high frequency linear US probe will be covered with a sterile sheath, and a 50 mm block needle will be used. The ultrasound probe will be placed vertically at the level of the L3 vertebra. After visualizing the guiding point spinous process and interspinal muscles, the probe will be moved laterally to visualize the longissimus and multifidus muscles. By using the in-plane technique, the block needle will be directed from medial to lateral, and after reaching the interfacial area between the longissimus and multifidus muscles, the block area will be confirmed by administering 5 ml of serum physiologically. Then, 20 ml of 0.25% local anesthetic will be administered. The same procedure will be applied to the other side. A total of 40 ml of local anesthetic solution will be used.
3. Postoperative analgesia management After anesthesia induction, 1 g iv Pracetamol before surgical incision and 20 mg iv Tenoxicam iv 20 mg 30 minutes before the end of the surgical procedure will be administered for postoperative analgesia. In the postoperative period, paracetamol 3x1 gr iv will be administered to the patients and iv Morphine infusion will be performed with a patient-controlled analgesia (PCA) device. By adding 0.5 mg/ml of morphine in the serum physiological, 1 mg bolus, 8 minutes lock time, and a maximum of 6 mg morphine per hour will be adjusted (12). Postoperative patient evaluation will be performed by another non-interventional anesthetist.

Postoperative pain assessment will be made using the NRS scoring (0 = no pain, 10 = most severe pain felt). Resting and mobile NRS scores will be recorded at 0, 2, 4, 8, 16, and 24 hours. NRS score < 4 will be targeted.

Sedation level will be monitored on a 4-point sedation scale (0=wake, eyes open, 1=sleepy but responds to verbal stimuli, 2=sleepy and difficult to awaken, 3=sleepy, cannot be woken by shaking).

Additional analgesic need, side effects such as nausea, vomiting, itching and complications that may occur due to block will be recorded.

References:

1. McGirt MJ et al. Recurrent disc herniation and long-term back pain after primary lumbar discectomy: review of outcomes reported for limited versus aggressive disc removal. Neurosurgery 2009; 64.2: 338-345.
2. Efthymiou CA, O'Regan DJ. Postdischarge complications: what exactly happens when the patient goes home?. Interactive cardiovascular and thoracic surgery 2011; 12.2: 130-134.
3. Benyamin R, Trescot AM, Datta S, et al. Opioid complications and side effects. Pain Physician 2008;11(2 Suppl l):S105.
4. Teddy PJ, Fabinyi G, Kerr JH, Briggs M. Bupivacaine infiltration after lumbar laminectomy: Local infiltration in the control of early postoperative lumbar laminectomy pain. Anaesthesia 1998;36(4): 380-383.
5. Dhanjal S, Tonder S. Quadratus Lumborum Block. 2020 Oct 23. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2020 Jan-. PMID: 30725897.
6. Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. PMID: 30688787.
7. Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID: 28154824; PMCID: PMC5244003.
8. Ueshima H, Otake H. Clinical experience of anterior quadratus lumborum block after lumber surgery. J Clin Anesth. 2017 Feb;37:131. doi: 10.1016/j.jclinane.2016.12.014. Epub 2017 Jan 9. PMID: 28235503.
9. Ueshima H, Hiroshi O. Lumbar vertebra surgery performed with a bilateral posterior quadratus lumborum block. J Clin Anesth. 2017 Sep;41:61. doi: 10.1016/j.jclinane.2017.06.012. Epub 2017 Jul 3. PMID: 28802611.
10. Hand WR et al. Thoracolum¬bar interfascial plane (TLIP) block: a pilot study in volunteers. Can J Anaesth 2015; 62: 1196-2000
11. Ueshima H et al. Efficacy of the thoracolumbar interfascial plane block for lumbar laminoplasty: a retrospective study. Asian spine journal 2017; 11.5: 722-725.
12. Gürkan Y et al. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. Journal of Clinical Anesthesia 50 (2018) 65-68

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old
2. ASA 1-2

Exclusion Criteria:

1. Bleeding diathesis
2. Opioid allergy
3. Infection in the area to be blocked
4. Have had previous lumbar surgery
5. Pregnant or suspected of pregnancy, breastfeeding
6. Gabapenthinoid, corticosteroid users
7. Those with kidney failure
8. Those with liver failure
9. Patients who cannot use a patient-controlled analgesia device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
postoperative analgesia | 24 hours
  Reducing the need for opioids used in the postoperative 24 hours in patients who have undergone lumbar spinal surgery

SECONDARY OUTCOMES:
opioid side effect | 24 hours
  To provide a lower postoperative pain score (NRS<4) in patients who have undergone lumbar spinal surgery, to reduce the risks of allergic reaction, nausea-vomiting, itching, sedation that may develop with opioid use.

CONTACTS AND LOCATIONS:
Locations (1):
- SAMSUN UNIVERSITY Samsun Training and research hospital, Samsun, Ilkadım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
After the work is completed

REFERENCES:
- [Background] Gurkan Y, Aksu C, Kus A, Yorukoglu UH, Kilic CT. Ultrasound guided erector spinae plane block reduces postoperative opioid consumption following breast surgery: A randomized controlled study. J Clin Anesth. 2018 Nov;50:65-68. doi: 10.1016/j.jclinane.2018.06.033. Epub 2018 Jul 2. PMID 29980005
- [Result] McGirt MJ, Ambrossi GL, Datoo G, Sciubba DM, Witham TF, Wolinsky JP, Gokaslan ZL, Bydon A. Recurrent disc herniation and long-term back pain after primary lumbar discectomy: review of outcomes reported for limited versus aggressive disc removal. Neurosurgery. 2009 Feb;64(2):338-44; discussion 344-5. doi: 10.1227/01.NEU.0000337574.58662.E2. PMID 19190461
- [Result] Efthymiou CA, O'Regan DJ. Postdischarge complications: what exactly happens when the patient goes home? Interact Cardiovasc Thorac Surg. 2011 Feb;12(2):130-4. doi: 10.1510/icvts.2010.249474. Epub 2010 Nov 30. PMID 21123196
- [Result] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Result] Teddy PJ, Fabinyi GC, Kerr JH, Briggs M. Bupivacaine infiltration after lumbar laminectomy. Local infiltration in the control of early postoperative lumbar laminectomy pain. Anaesthesia. 1981 Apr;36(4):380-3. doi: 10.1111/j.1365-2044.1981.tb10242.x. PMID 7018317
- [Result] Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. No abstract available. PMID 30688787
- [Result] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Result] Ueshima H, Otake H. RETRACTED: Clinical experience of anterior quadratus lumborum block after lumber surgery. J Clin Anesth. 2017 Feb;37:131. doi: 10.1016/j.jclinane.2016.12.014. Epub 2017 Jan 9. No abstract available. PMID 28235503 (Retraction: PMID 35393201 J Clin Anesth. 2022 Aug;79:110740)
- [Result] Ueshima H, Hiroshi O. RETRACTED: Lumbar vertebra surgery performed with a bilateral posterior quadratus lumborum block. J Clin Anesth. 2017 Sep;41:61. doi: 10.1016/j.jclinane.2017.06.012. Epub 2017 Jul 3. No abstract available. PMID 28802611 (Retraction: PMID 35396108 J Clin Anesth. 2022 Aug;79:110790)
- [Result] Hand WR, Taylor JM, Harvey NR, Epperson TI, Gunselman RJ, Bolin ED, Whiteley J. Thoracolumbar interfascial plane (TLIP) block: a pilot study in volunteers. Can J Anaesth. 2015 Nov;62(11):1196-200. doi: 10.1007/s12630-015-0431-y. Epub 2015 Jul 7. PMID 26149600
- [Result] Ueshima H, Ozawa T, Toyone T, Otake H. Efficacy of the Thoracolumbar Interfascial Plane Block for Lumbar Laminoplasty: A Retrospective Study. Asian Spine J. 2017 Oct;11(5):722-725. doi: 10.4184/asj.2017.11.5.722. Epub 2017 Oct 11. PMID 29093781